CLINICAL TRIAL: NCT00948883
Title: Epidemiological, Immunological, Pathological and Pharmacogenetic Study of Cancers Occuring After Solid Organs Transplants
Brief Title: Study of Cancers After Solid Organs Transplants
Acronym: K-GREF
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: CANCEROPOLE Ile-de-France (Unknown)
Responsible Party: Sponsor
Other Study IDs: DRCD CANC 0701
Record Dates: First submitted 2009-07-28; First posted 2009-07-29 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-04

CONDITIONS: Cancer; Organ Transplantation
Keywords: organ transplant; cancer; biobank; immunosuppressive drugs; lymphoma
MeSH Terms: conditions — Neoplasms; Lymphoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, frozen tissue
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Patient-Case: Transplanted patient with cancer
- Patient-Control: Transplanted patient without cancer

SUMMARY:
About 1500 solid organs transplants are performed each year in the Paris agglomeration.

Cancer risk in the transplanted is about three times higher than in a population of the same age without any organ transplant. Thus cancer is an important problem for organ transplant.

These cancers can be related to many factors :

* Post-transplant cancers are due in part to the non specific immunosuppression, which leads to oncogenic viruses replication, and then produces virus inducted cancers (as lymphoma due to EBV virus).
* Post-transplant cancers can also be due to the carcinogenic factors of the immunosuppressive drugs (as cyclosporine or tacrolimus, which can cause the appearance of metastases). However, a new type of immunosuppressive drugs (mTOR inhibitors) appear to have anti-cancer properties.
* Post-transplant cancers which are not virus-inducted can be relied to genetic factors of the transplanted patient and/or the transplant donor.

There are 4 axes in this study :

* Axis 1 : Epidemiological, clinical and biological study of the incident cancers in transplanted patients.
* Axis 2 : Qualitative and quantitative immunological study of lymphocyte cells by the transplanted patient (determine their characteristics when a cancer appears).
* Axis 3 : Pathological and genetic study of the post-transplant cancer cells (see if the cancer is caused by the donor or the recipient). Creation of a biobank.
* Axis 4 : Pharmacogenetic study of the immunosuppressive drugs (determine the impact of patient genetic variability on tolerance and efficiency of the immunosuppressive drugs).

DETAILED DESCRIPTION:
This is an observational and comparative study (2 control patients are recruited for each 1 case patient).

A case patient is a patient who has developed a cancer after his/her transplant.

A control patient is a patient who has not developed a cancer after his/her transplant.

These 2 groups will be matched according to specific inclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman after 18 years old
* Transplanted with a solid organ (heart, kidney, lung,liver)
* Informed Consent Form signed
* For the patients-case: Patients who developed a post-transplant cancer
* For the patients-control: Patients who didn't develop a post-transplant cancer

Exclusion Criteria:

* Cancer as transplant indication ( except liver )
* HIV positive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with solid organ transplant who have developed a cancer. Patients with solid organ transplant who have not developed a cancer.
Sampling Method: Non-Probability Sample
Enrollment: 330 (Actual)
Dates: Start 2008-10; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Incidence of cancer among transplanted patients. | At the day of blood collection

SECONDARY OUTCOMES:
Characteristics of the tumors. | At the day of blood collection
Risk factors of the tumors. | At the day of blood collection

CONTACTS AND LOCATIONS:
Overall Officials: Michel MARTY, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Bicêtre - Assistance Publique-Hôpitaux de Paris, Le Kremlin-Bicêtre, France